CLINICAL TRIAL: NCT05938153
Title: Evaluation of Metabolic Syndrome, Frailty, Locomotive Syndrome, Balance and Physical Fitness in Elderly Individuals
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Alper Kemal Gürbüz, research asistant, Kırıkkale University
Other Study IDs: Gurbuz02
Record Dates: First submitted 2023-07-03; First posted 2023-07-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2023-07

CONDITIONS: Geriatrics; Fragility; Locomotor; Physical Fitness; Balance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- geriatrics individuals
  Interventions: Other: observational physical tests

INTERVENTIONS:
Other: observational physical tests — Geriatric Locomotive Function Scale:
  This scale consists of a questionnaire of 25 items that can be easily understood by the elderly and each item is graded between 0 and 4 points. The total score is the result of the sum of all items ranging from 0 to 100; the higher the score, the higher the physical impairment of the elderly, with a score of 16 being the cut-off point for locomotive syndrome. The GLFS-25 includes 4 questions about pain, 16 questions about activities of daily living, 3 questions about social performance and 2 questions about mental health status to assess geriatric individuals. Turkish validity and reliability of the questionnaire was conducted by Sadikoglu.

SUMMARY:
Metabolic syndrome (MetS) or syndrome X, which is increasingly prevalent in the world and in our country, is a disease that includes abdominal obesity, dyslipidemia, impaired glycemic control and hypertension components. It causes cardiovascular events such as myocardial hypertrophy, left ventricular diastolic dysfunction, atrial dilatation and atrial fibrillation. Low levels of physical activity can be caused by a wide variety of factors including environmental and genetic factors, age, race, sarcopenia, poor eating habits, postmenopausal period and smoking history. Factors such as genetic differences, diet, physical activity, age, gender and eating habits are reported to affect the prevalence of (MetS) and its components. Frailty is also emerging as a major issue for the elderly due to its debilitating effects on health outcomes. Frailty is a geriatric syndrome characterized by a gradual decrease in homeostatic tolerance and physiological reserve following exposure to stressors. Frailty predisposes older people to falls, delirium, hospitalizations and even death and is therefore considered a crucial transition between healthy ageing and disability. As a result of aging, degenerative changes in the central and peripheral vestibular system have been found. With age, the ability to regulate movement is impaired as a result of insufficient information in any of the sensory receptors or any disorder affecting the processing of these messages. This directly affects balance and postural control, leading to an increased risk of falls. In the light of the results of the studies in the literature, degenerative changes are observed in many systems in geriatric individuals and while the incidence of metabolic syndrome in these individuals is high, the number of studies evaluating their effects is not sufficient. Based on these deficiencies, it is aimed to examine metabolic syndrome, frailty, locomotive syndrome, balance and physical fitness in elderly individuals.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 and over,
* Volunteering to participate in the research
* No cooperation and communication problems

Exclusion Criteria:

* Individuals with neurological and orthopedic problems
* Uncontrolled hypertension
* Those with cardiac disorders
* Those with cooperation and communication problems

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Individuals aged 65 and over, 10 individuals
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Geriatric Locomotive Function Scale: | 10 minute
  This scale consists of a questionnaire of 25 items that can be easily understood by the elderly and each item is graded between 0 and 4 points. The total score is the result of the sum of all items ranging from 0 to 100; the higher the score, the higher the physical impairment of the elderly, with a score of 16 being the cut-off point for locomotive syndrome. The GLFS-25 includes 4 questions about pain, 16 questions about activities of daily living, 3 questions about social performance and 2 questions about mental health status to assess geriatric individuals. Turkish validity and reliability of the questionnaire was conducted by Sadikoglu.

SECONDARY OUTCOMES:
Chair sit-lie test | 5 minute
  The patient is asked to sit and stand as quickly as possible in a chair with a seat height of 43.2 cm and a supported back. The patient sits on the chair.He crosses his hands on his chest. 2 attempts are made before the test. A stopwatch is kept for 30 seconds and the number of sit-ups is noted. Less than 10 sit-ups in 30 seconds indicates lower extremity muscle weakness
Two-minute step test | 2 minute
  It is applied to evaluate aerobic endurance. In order to perform the test correctly, the distance at which the participant will lift the knee is determined as the midpoint between the knee joint and the crista iliaca and marked on the wall. For a better understanding of the test is demonstrated practically. The participant is asked to start with the right foot and rhythmically raise their feet to the marked height for 2 minutes. The number of standardized right steps repeated for two minutes is recorded as a score.
Weight lifting test | 2 minute
  It is applied to evaluate upper extremity muscle strength. Participant's feet is asked to sit towards the side of the chair while on the floor. The participant is asked to bend and extend their arms by lifting the dumbbell with the given instruction. As weight dumbbells of 3.63 kg for men (8-lb) and 2.27 kg for women (5-lb) are used. For a better understanding of the test, it was demonstrated and practiced. In the test, the maximum possible number of repetitions performed with the dominant arm for 30 s is considered as the score.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Kırıkkale, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No